CLINICAL TRIAL: NCT05020834
Title: Effect of Functional Electrical Stimulation Versus TheraTogs on Gait and Balance in Children With Hemiplegic Cerebral Palsy
Brief Title: Effect of Functional Electrical Stimulation Versus TheraTogs on Treatment of Children With Hemiplegic Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm Al-Qura
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Electrical Stimulation Group (Experimental): Functional Electrical Stimulation Group received 1.5 hours of conventional physical therapy program /session - 3 sessions weekly - three successive months + 1/2 hour of the gait training program with functional electrical stimulation /session - 3 sessions weekly - three successive months.
  Interventions: Other: Functional Electrical Stimulation
- TheraTogs Group (Experimental): TheraTogs Arm The participating children will wear TheraTogs orthotic undergarment and strapping as preparatory stage without application of any exercise program with gradually increasing the worn time till reaching the 8 hours per day.
  Interventions: Other: TheraTogs Orthotic Undergarment

INTERVENTIONS:
Other: Functional Electrical Stimulation — Functional Electrical Stimulation Group received 1.5 hours of conventional physical therapy program /session - 3 sessions weekly - three successive months + 1/2 hour of the gait training program with functional electrical stimulation /session - 3 sessions weekly - three successive months.
  Arms: Functional Electrical Stimulation Group
Other: TheraTogs Orthotic Undergarment — TheraTogs Arm The participating children worn TheraTogs orthotic undergarment and strapping as preparatory stage without application of any exercise program with gradually increasing the worn time till reaching the 8 hours per day.
  Arms: TheraTogs Group

SUMMARY:
To compare the effect of functional electrical stimulation (FES) versus TheraTogs on Gait and Balance in children with hemiplegic CP.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of FES versus TheraTogs on Gait and Balance in children with hemiplegic CP. Thirty children with hemiplegic CP will be assigned randomly into two groups (A & B). Group A received FES by using the WalkAide foot drop stimulator while group B received TheraTogs. Patients' evaluation will be carried out before and after training to assess gait and balance performance.

ELIGIBILITY:
Inclusion Criteria:

* Their weight should be less than 40 kg.
* The spasticity degrees of the affected lower limb will range between grades (1, 1+ & 2) according to Modified Ashworth Scale (MAS).
* Those children functioning scores at Gross Motor Function Classification System (GMFCS) Levels I and II.
* They can walk 10 min conditionally without an orthosis.
* Ought to be intellectually skilled and ready to comprehend and take after directions.
* They will have neither serious nor recurring medical complications.
* Children's height will be more than 100 cm to fit with the Biodex balance equipment that will be used in this study to evaluate balance performance.
* No serious hip & knee flexion tightness will be present. Knee flexion at starting contact should be between 20-40º .
* Peroneal nerve and the proximal leg muscles ought to be in place.
* They ought to have no significant issues influencing balance other than spasticity.

Exclusion Criteria:

* Children who demonstrate skin diseases or allergic reactions to adhesive tape or any other materials used in this study.
* Children with visual, auditory or perceptual deficits.
* Children with surgical interference for the lower limb.
* Children with seizures or epilepsy.
* Children who received botulinum toxin in the lower extremity musculature during the past 6 months or who wish to receive it within the period of study, other spasticity medication within 3 months of pre-treatment testing .
* Children with pacemakers or other diseases that are contraindicated by electrical stimulation.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline spatial and temporal gait parameters at 3 months | Baseline and 3 months post-intervention
  Gait parameters were evaluated for every child at baseline and 3 months post-intervention using the Pro-Reflex motion analysis system (Qualisys; Qualisys Inc, Goeteborg, Sweden). For the purpose of this study four commonly used and reliable gait parameters were examined: stride length, step length, velocity, cadence, and stance and swing phase percentage.
Change from baseline postural stability at 3 months | Baseline and 3 months post-intervention
  Postural stability were evaluated at baseline and 3 months post-intervention using the Biodex Balance System (BBS) (Balance System SD, Shirely, NY, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M Elshamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Maternity and Children Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No